CLINICAL TRIAL: NCT03666585
Title: Comparison of the Accuracy in Rehabilitation Exercise Between Mobile Application Actuated Rehabilitation Exercise Guidance and Routine Rehabilitation Exercise Guidance for the Primary Osteoarthritis Knee Patients : A Randomized Controlled Trial
Brief Title: Comparison of the Accuracy in Rehabilitation Exercise Between Mobile Application Actuated Rehabilitation Exercise Guidance and Routine Rehabilitation Exercise Guidance for the Primary Osteoarthritis Knee Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Satit Thiengwittayaporn, Associate Professor, Navamindradhiraj University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COA 034/2561
Record Dates: First submitted 2018-09-03; First posted 2018-09-12 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Mobile Application Actuated Rehabilitation Exercise Guidance; Routine Rehabilitation Exercise Guidance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile application actuated rehabilitation exercise guidance (Active Comparator)
  Interventions: Other: mobile application actuated rehabilitation exercise guidance
- routine rehabilitation exercise guidance (Active Comparator)
  Interventions: Other: routine rehabilitation exercise guidance

INTERVENTIONS:
Other: mobile application actuated rehabilitation exercise guidance — Mobile applications (also known as mobile apps) are software programs developed for mobile devices such as smartphones and tablets, to teach full function following injury and involves restoring strength, flexibility, endurance, and power.
  Arms: mobile application actuated rehabilitation exercise guidance
Other: routine rehabilitation exercise guidance — the teach to practice full function following injury and involves restoring strength, flexibility, endurance, and power. It is achieved through various exercises and drills
  Arms: routine rehabilitation exercise guidance

SUMMARY:
Evaluate the accuracy of physical therapy in various positions after 4 weeks of training, comparison of the accuracy in rehabilitation exercise between mobile application actuated rehabilitation exercise guidance and routine rehabilitation exercise guidance for the primary osteoarthritis knee patients

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of knee
* Have an android phone and use the application

Exclusion Criteria:

* There are other complications that may affect physiotherapy
* Communication problems
* Has been trained in physical therapy for osteoarthritis patients
* Have had total knee arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Outcome measurement to compare the accuracy | 1 month
  To measurement by number of patient performing correct exercise has 3 exercise 10 steps and number of patient performing incorrect exercise has 3 exercise 10 steps. to compare the accuracy when osteoarthritis knee patients do rehabilitation using mobile application actuated rehabilitation exercise guidance and routine rehabilitation exercise guidance.If the patient is able to perform at least 8 times (80%), the patient will be define as corrected physical therapy, We compare the correction of physical therapy between the groups.
Patient satisfaction of rehabilitation method | 1 month
  To compare the satisfaction of rehabilitation method after rehabilitation program of physical therapy by questionnaire. The satisfaction score has 5 point.
  The 1 point mean the least satisfaction of patient to the method. The 2 point mean the less satisfaction of patient to the method. The 3 point mean the moderate satisfaction of patient to the method. The 4 point mean the much satisfaction of patient to the method. The 5 point mean the most satisfaction of patient to the method.

CONTACTS AND LOCATIONS:
Overall Officials: Satit Thiengwittayaporn, M.D., Principal Investigator — Department of Orthopaedics, Faculty of Medicine Vajira Hospital, Navamindradhiraj University
Locations (1):
- Navamindradhiraj University, Dusit, Bangkok, Thailand

REFERENCES:
- [Derived] Thiengwittayaporn S, Wattanapreechanon P, Sakon P, Peethong A, Ratisoontorn N, Charoenphandhu N, Charoensiriwath S. Development of a mobile application to improve exercise accuracy and quality of life in knee osteoarthritis patients: a randomized controlled trial. Arch Orthop Trauma Surg. 2023 Feb;143(2):729-738. doi: 10.1007/s00402-021-04149-8. Epub 2021 Aug 28. PMID 34453570